CLINICAL TRIAL: NCT04078828
Title: Pelvic Floor Reconstruction (PR) in Endoscopic Low Anterior Resection for Rectal Cancer
Brief Title: PR in Endoscopic LAR for Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Li Chuan, Secretary of General Surgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRLAR-SURGERY
Record Dates: First submitted 2019-08-15; First posted 2019-09-06 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Rectal Carcinoma
Keywords: minimally invasive surgical
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR (Active Comparator)
  Interventions: Procedure: Pelvic floor Reconstruction
- Non-PR (Active Comparator)
  Interventions: Procedure: Pelvic floor Reconstruction

INTERVENTIONS:
Procedure: Pelvic floor Reconstruction — Pelvic floor Reconstruction after laparoscopic anterior resection and double-stapling technique anastomosis were finished.

SUMMARY:
The anastomotic leakage remains the major early complication after laparoscopic anterior resection(LAR) for medium & low rectal cancer. Pelvic floor reconstruction (PR) is a key step in various standard resections for open radical rectal cancer surgery, which was considered to be helpful for decreasing the rate of leakage. However, PR in endoscopic LAR surgery is not routine practice and remains controversial. The purpose of this study is to evaluate the efficacy of PR during LAR for mid/low rectal carcinoma, especially in preventing anastomotic leakage.

DETAILED DESCRIPTION:
Eligible patients with rectal cancer will be randomly assigned to group with pelvic floor reconstruction(PR) versus group without pelvic floor reconstruction(NPR).

We want to investigate the rate of anastomotic leakage and re-operation between the two groups, some other relevant outcomes will be concerned all the same.

ELIGIBILITY:
Inclusion Criteria:

1. patients with histologically proven rectal adenocarcinoma
2. tumor located in the middle and lower rectum and anastomosis under the peritoneal reflection
3. Tumor assessed as a depth of invasion that was confined to pT1-pT3, bN0-1M0 by ultrasound colonoscopy and/or pelvic MRI
4. Negative circumferential resection margin confirmed by MRI
5. Performance status (ECOG) 0~1
6. Written informed consent for participation in the trial

Exclusion Criteria:

1. History of accepting lower abdominal surgery.
2. More than one colorectal tumor
3. Patients with unresectable distant metastasis or multiple metastases
4. Received neoadjuvant radiotherapy before surgery
5. Signs of acute intestinal obstruction, bleeding or perforation needing emergency surgery
6. Patients and/or family members cannot understand and accept this study
7. Non-rectal adenocarcinoma was confirmed by postoperative pathological examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The rate of anastomotic leakage after laparoscopic anterior resection for rectal cancer | 30 days after surgery
Re-operation rate after anastomotic leakage | 30 days after surgery
The rate of general complications | 30 days after surgery

SECONDARY OUTCOMES:
Operative time | Operation day
Postoperative hospital stay | 1 year after surgery
Incidence of defecation dysfunction | From the date of operation until the date of complication,assessed up to 3 years
3-year local recurrence rate | From date of operation until the date of local-recurrence (up to 3 years)
5-year disease-free survival | From date of operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Postoperative quality of life as assessed by EORTC QLQ-C30 questionnaire | 1 year after operation
Blood loss | Operation day
White blood cells(WBC) ,C-reactive protein (CRP) and procalcitonin (PCT) count in the blood sample | 1 days after surgery
White blood cells(WBC) ,C-reactive protein (CRP) and procalcitonin (PCT) count in the blood sample | 3 days after surgery
White blood cells(WBC) ,C-reactive protein (CRP) and procalcitonin (PCT) count in the blood sample | 5 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Center of PLA, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided